CLINICAL TRIAL: NCT02801175
Title: Differential Effect of Radiofrequency and Cryoballoon Ablation on Left Atrial Appendage Emptying Flow Velocity
Brief Title: Effect of Left Atrial Ablation on Left Atrial Appendage Emptying Flow Velocity
Acronym: ABLAA-FV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: G.Gennimatas General Hospital (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Associate Professor of Cardiology, National and Kapodistrian University of Athens
Other Study IDs: 1/13.6.2016
Record Dates: First submitted 2016-06-13; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- RF: Patients with paroxysmal atrial fibrillation slated for radiofrequency pulmonary vein isolation
  Interventions: Procedure: Pulmonary vein isolation
- Cryoballoon: Patients with paroxysmal atrial fibrillation slated for cryoballoon pulmonary vein isolation
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation

SUMMARY:
Consecutive patients with paroxysmal AFib scheduled to undergo pulmonary vein isolation either with radiofrequency (RF) or cryoballoon will be included. Left atrial appendage emptying flow velocity (LAA-EFV) will be measured with transesophageal echocardiography (TEE) immediately before and following left atrial ablation (1 month post). The change in LAA-EFV will be compared between the two groups (RF versus Cryo).

ELIGIBILITY:
Inclusion Criteria:

Paroxysmal atrial fibrillation, no absolute contraindication for anticoagulation

Exclusion Criteria:

Previous cardiac surgery Previous left atrial ablation History of cerebrovascular event Presence of LAA thrombus Inability to provide informed consent

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ablation-naive patients with paroxysmal AFib
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
LAA-EFV | 1 month
  Left atrial appendage emptying flow velocity

SECONDARY OUTCOMES:
LAA-EFV | 3 months
  Left atrial appendage emptying flow velocity

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Dept. of Cardiology, Univ of Athens Med Sch, Athens, Greece